CLINICAL TRIAL: NCT05304546
Title: Overcoming Primary Resistance to Immunotherapy in Metastatic Melanoma Patients by Transient Addition of BRAF and MEK Inhibitors Followed by Pembrolizumab: A Pivotal Open Label, Single-site Study
Brief Title: Overcoming Primary Resistance to Immunotherapy in Metastatic Melanoma
Acronym: MK3475-C01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Ronnie Shapira (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Ronnie Shapira, Head of the Ella Lemelbaum Institute for Immuno-Oncology, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9222-22-SMC
Record Dates: First submitted 2022-03-16; First posted 2022-03-31 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Malignant Melanoma; Metastatic Melanoma; Immunotherapy; BRAF V600E; Malignant Melanoma Stage IV
Keywords: Melanoma; Primary Resistance to Immunotherapy; Neoplasm
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — pembrolizumab; encorafenib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm MK3475, encorafenib and binimetinib (Experimental): Intravenous pembrolizumab 400 mg Q6W + oral encorafenib 450 mg QD + oral binimetinib 45mg BID, for the first 4 weeks of the study. Starting week 5, monotherapy pembrolizumab 400 mg Q6W.
  Interventions: Drug: Pembrolizumab; Drug: Encorafenib; Drug: Binimetinib

INTERVENTIONS:
Drug: Pembrolizumab — Solution for IV
  Other Names: Keytruda; MK3475
Drug: Encorafenib — Oral QD
  Other Names: Braftovi
Drug: Binimetinib — Oral BID
  Other Names: Mektovi

SUMMARY:
This study will enroll metastatic (Stage IV or inoperable stage III) melanoma (MM) patients carrying a BRAF V600E/K mutation with confirmed primary resistance to standard of care immunotherapy (single agent PD-1 or a combination of CTLA-4/PD-1 blockade). Patients must be naïve to therapy with BRAF+MEK inhibitors, with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

DETAILED DESCRIPTION:
Treatment groups (single-arm):

During Weeks 1-4 of the study, subjects will receive intravenous pembrolizumab 400 mg every 6 weeks (Q6W), oral encorafenib 450 mg once daily and oral binimetinib 45mg twice daily. From Week 5-13, participants will receive intravenous pembrolizumab 400 mg every 6 weeks. From Week 13 to 2 years, subjects with a response of stable disease or better (determined by CT every 3 months) will receive pembrolizumab 400mg Q6W until evident progressive disease by Response Evaluation Criteria In Solid Tumors (RECIST), unacceptable toxicity, withdrawal of consent, or until completion of 17 treatment cycles (approximately 2 years) with pembrolizumab.

Participants who stop study treatment after receiving 17 administrations of pembrolizumab for reasons other than disease progression or intolerability, or participants who attain a complete response (CR) and stop study treatment may be eligible for up to 1 year of treatment with pembrolizumab (~8 cycles) upon experiencing disease progression (Second Course Phase).

Tumor biopsies and blood (peripheral blood mononuclear cells [PMBC] and plasma) will be obtained upon patient recruitment, during the screening period, after 4 weeks of treatment and at 13 weeks.

Primary Translational Objectives & Hypothesis:

1. To determine the decrease in nuclear c-MYC levels in situ in tumor biopsies and blood following treatment.
2. To determine the increase in mitochondrial activity protein profile (Acetyl-CoA acetyltransferase [ACAT1] and Hydroxyacyl-CoA dehydrogenase trifunctional multienzyme complex subunit alpha [HADHA]) in the tumor cells1 in situ following treatment.
3. To determine the increase in CD8+ counts in situ following treatment. Hypothesis: c-MYC impairs interferon gamma (IFNγ) responsiveness and drives anaerobic metabolism,which reduces antigenicity. MAPK activation through the BRAF V600 mutation leads to c-MYC activation and its nuclear translocation in MM patients, directly inhibiting aerobic metabolism in melanoma cells in-vitro. Thus, BRAF V600 seems to drive both mechanisms #1 and #2, highlighting its potential targeting to revert primary immune resistance.

The investigators hypothesize that BRAF inhibition will deactivate c-MYC and drive tumor cell metabolism towards oxidative phosphorylation. c-MYC deactivation is expected to alleviate IFNγ resistance. Aerobic metabolism of tumor cells is expected to increase their immunogenicity. The combined effect is expected to overcome primary resistance and reinvigorate local immune response. This is expected to be evident by increased T cell influx, which is associated with successful checkpoint inhibition, and could be further perpetuated with PD-1 blockade.

Primary Clinical Objectives & Hypothesis:

To determine the best overall response rate (BORR) to pembrolizumab. Hypothesis: The immunological alteration in the tumor and its microenvironment will provide the grounds for pembrolizumab to induce a clinical response.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of metastatic melanoma with BRAF V600E/K mutation will be enrolled in this study.
2. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 125 days (5 terminal half-lives for pembrolizumab) after the last dose of study treatment and refrain from donating sperm during this period.
3. Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
4. Participants must have progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:

   1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb. Note: participants who have received prior anti-PD-1+ CTLA4 may be included in the study.
   2. The last line prior to inclusion in the study must include an approved anti-PD-1 therapy.
   3. Has demonstrated clinical PD after anti-PD-1/L1 The initial evidence of PD is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented PD, in the absence of rapid clinical progression.
   4. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.
   5. This determination is made by the investigator. Once PD is confirmed, the initial date of PD documentation will be considered the date of disease progression.
5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
6. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Have not been previously treated with BRAF inhibitors and/or MEK inhibitors.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of treatment initiation.
9. Have adequate organ function as defined below. Specimens must be collected within 10 days prior to the start of study treatment.

Adequate Organ Function Laboratory Values:

Absolute neutrophil count (ANC) ≥1500/μL Platelets ≥100 000/μL Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La Creatinine OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases) Coagulation: International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment initiation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior systemic anti-cancer therapy including investigational agents within 2 weeks prior to treatment initiation.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

   Note: If the participant had major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
3. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
4. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
5. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.

   Note: This time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers
8. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
9. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
11. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a known history of Human Immunodeficiency Virus (HIV) infection.
14. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus infection (defined as detected HCV RNA [qualitative]).
15. Has a known history of active Bacillus Tuberculosis (TB).
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
19. Has had an allogenic tissue/solid organ transplant.
20. Baseline ejection fraction <50%, or below the institutional lower limit of normal (LLN).
21. A history of retinal vein occlusion (RVO) or current risk factors for RVO including uncontrolled glaucoma or a history of hyperviscosity or hypercoagulability syndromes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Decrease in nuclear c-MYC levels in situ by 50% | 48 months
  Results of IHC with readout of intensity and percentage with nuclear localization will be used to evaluate this outcome. C-MYC will be evaluated on the basis of intensity (0 to +3).
Increase in mitochondrial proteins ACAT1 and HADHA in the tumor cells in situ by 50% | 48 months
  HADHA and ACAT1 will be evaluated on the basis of intensity (0 to +3) and percentage of positive cells
Increase in CD8+ counts in situ by 50% | 48 months
  Results of IHC enabling CD8 counts will be used to evaluate this outcome
Best overall response rate (BORR) to pembrolizumab | 48 months
  Assessed by RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 48 months
  Assessed by RECIST 1.1
Duration of response (DoR) | 48 months
  Assessed by RECIST 1.1
Response rate to targeted therapy upon progression | 48 months
  Assessed by RECIST 1.1
Number of participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | 48 months
  Safety and tolerability of the investigational medicinal products

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Shapira-Frommer, Dr, Principal Investigator — Ella Lemelbaum Institute for Immuno-Oncology & Melanoma, Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel, Israel

IPD SHARING:
Plan to Share IPD: No